CLINICAL TRIAL: NCT03684499
Title: Role of Fluid Supplementation in Neonatal Unconjugated Hyperbilirubinemia
Brief Title: Fluid in Neonatal Hyperbilirubinemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasmeen Hasaneen Mohamed, role of fluid supplementation in neonatal unconjugated hyperbilirubinemia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: fsnh
Record Dates: First submitted 2018-09-20; First posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Bilirubinemia
MeSH Terms: conditions — Hyperbilirubinemia | interventions — Phototherapy; Lactation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (1) (Other): The subjects will be divided into two equal groups Study group and control group by randomization. The study group will be given IV fluid supplementation with 0.5% normal saline in dextrose 5%for period of 24hours . The volume of supplementation included a presumed deficit of 50 ml/kg (equivalent to mild dehydration), half of daily maintenance fluid for 24 hours in accordance to standard norms and extra 20 ml/kg per day as a phototherapy allowance. In addition, they will continue breastfeeding. The control group will be continued on breast feeding , before the randomization procedure. All the infants will get phototherapy by standard method. Phototherapy will be discontinued when the bilirubin level will be <15 mg/dl.
  Interventions: Other: fluid supplementation; Other: breast feeding
- control group( 2) (No Intervention): The subjects will be divided into two equal groups Study group and control group by randomization. The study group will be given IV fluid supplementation with 0.5% normal saline in dextrose 5%for period of 24hours . The volume of supplementation included a presumed deficit of 50 ml/kg (equivalent to mild dehydration), half of daily maintenance fluid for 24 hours in accordance to standard norms and extra 20 ml/kg per day as a phototherapy allowance. In addition, they will continue breastfeeding. The control group will be continued on breast feeding , before the randomization procedure. All the infants will get phototherapy by standard method. Phototherapy will be discontinued when the bilirubin level will be <15 mg/dl.

INTERVENTIONS:
Other: fluid supplementation — The subjects will be divided into two equal groups Study group and control group by randomization. The study group will be given IV fluid supplementation with 0.5% normal saline in dextrose 5%for period of 24hours . The volume of supplementation included a presumed deficit of 50 ml/kg (equivalent to mild dehydration), half of daily maintenance fluid for 24 hours in accordance to standard norms and extra 20 ml/kg per day as a phototherapy allowance. In addition, they will continue breastfeeding. All the infants will get phototherapy by standard method. Phototherapy will be discontinued when the bilirubin level will be <15 mg/dl.
  Other Names: phototherapy
  Arms: study group (1)
Other: breast feeding — The subjects will be divided into two equal groups Study group and control group by randomization . The control group will be continued on breast feeding , before the randomization procedure. All the infants will get phototherapy by standard method. Phototherapy will be discontinued when the bilirubin level will be <15 mg/dl.(Bandyopadhyay et al, 2017)
  Arms: study group (1)

SUMMARY:
Hyperbilirubinemia is a common neonatal problem. bilirubin is potentially toxic to central nervous system and can cause serious permanent complication called kernicterus, in which brain stem nuclei and basal ganglia are damaged,resulting in cerebral palsy.In Hyperbiliubinemia,rapid reduction of serum bilirubin level is of utmost importance.

Two commonly used mode of therapy are phototherapy and exchange transfusion. Phototherapy has some side effects such as diarrhea, skin rash, dehydration, overheating, mother-baby bonding disruption.On the other hand, complication of exchange transfusion include infections, emboli,anemia,apnea and hypocalcemia.

while IV fluid supplementationis postulated to decrease bilirubin concentration directly through a reduction of haemoconcentration, increasing enteral feed volume is proposed to decrease bilirubin concentration through reduced enterohepatic circulation via an increased gut peristalsis.

DETAILED DESCRIPTION:
Bilirubin encephalopathy or kernicterus Unconjugated bilirubin is lipid soluble and therefore can cross the blood brain barrier .There it can deposit in areas of the brain, with a predilection for deposition in the basal ganglia, auditory pathways, and oculomotor nucleus. This deposition and accompanying damage result in the classical symptoms associated with kernicterus. Hypoxia, acidosis, prematurity, and genetic predispositions all increase the risk for kernicterus.In well term babies risk for kernicterus increases after bilirubin levels cross (20 mg/dL) and it is very high above (30 mg/dL). In preterm babies the threshold for damage from bilirubin could be as low as(20mg/dl). The risk increases with increasing serum levels of unconjugated bilirubin.

Acute bilirubin encephalopathy presents as lethargy, high pitched cry, poor feeding, abnormal tone, opisthotonus, upgaze palsy and seizures. Aggressive treatment at this stage can reduce the damage caused. Chronic bilirubin encephalopathy leads to conditions like choreoathetoid cerebral palsy, high frequency hearing loss, dental dysplasias and oculomotor palsies.

ELIGIBILITY:
Inclusion Criteria:

1 -Ful term ,Body weight (≥2.5kg). 2- total serum bilirubin range(≥18mg/dl to≤25mg/dl). 3-Non -haemolytic type of jaundice. 4-Ratio of conjugated bilirubin :unconjugated bilirubin is 1:5

Exclusion Criteria:

1 - Body weight ≤2.5kg. 2- Evidence of haemolysis. 3- Obvious features of dehydration. 4- Major congenital malformation . 5- Baby received already IV fluid for any reason. 6- Septicemia . 7-GIT functional or organic obstruction .

Ages: 3 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
decrease of bilirubin level after fluid supplementation | 24 hours
  bilirubin level will be measured on admission and after 24 hours and

SECONDARY OUTCOMES:
phototherapy | 24
  reduce duration of phototherapy

CONTACTS AND LOCATIONS:
Overall Officials: Yasmeen Hasaneen, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided